CLINICAL TRIAL: NCT06227572
Title: Cognition After Obstructive Sleep Apnea (OSA) Treatment Among Native American People (CATNAP)
Brief Title: Cognition After OSA Treatment Among Native American People (CATNAP)
Acronym: CATNAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Missouri Breaks Industries Research, Inc. (Other); University of Washington (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Denise Dillard, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01AG066584 (NIH)
Record Dates: First submitted 2022-02-23; First posted 2024-01-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Cognitive Change
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The CATNAP MI intervention consists of 3 Motivational Interviewing sessions to address obstructive sleep apnea (OSA), positive airway pressure (PAP) adherence, and risk of Alzheimer's disease and related dementias (ADRD) in American Indians and electronic messaging to support PAP adherence, and usual care. Data will be collected at baseline, 3-months, and 9-months.
  Interventions: Behavioral: CATNAP MI
- Waitlist Control Group (No Intervention): Usual care, consisting of an in-service on how to operate the PAP machine, and a mask fitting to select the most comfortable, effective mask for the individual. After 4-6 weeks of use, the participant will be contacted by Missouri Breaks Durable Medical Equipment to review objective adherence data and address any challenges or barriers to therapy such as treatment-emergent central apneas. Data will be collected at baseline, 3-months, and 9-months.

INTERVENTIONS:
Behavioral: CATNAP MI — Three motivational interviewing (MI) sessions will be facilitated by trained MI staff and will focus on improving participants' knowledge about their OSA diagnosis, understanding of sleep health, and increasing PAP use. Sessions will also provide information about health benefits associated with good sleep and will help participants create an action plan regarding their PAP use and indicators of success, when appropriate.
  Electronic messaging will be standardized for frequency and content but personalized to participants' preferred mode of delivery. Messages will focus on PAP adherence or non-adherence.
  Arms: Intervention Group

SUMMARY:
This research project will develop and implement a motivational interviewing and electronic messaging intervention to address obstructive sleep apnea (OSA), positive airway pressure (PAP) adherence, and risk of Alzheimer's disease and related dementias in American Indians. The project will work with American Indian Elders, aged 50 years and older, from three Northern Plains Reservations and surrounding communities. A total of 300 American Indian elders with a confirmed OSA diagnosis and prescribed PAP therapy will be randomized to receive usual care consisting of PAP therapy alone (control condition) or usual care plus the culturally informed CATNAP MI component (intervention condition).

DETAILED DESCRIPTION:
The investigators will develop a multilevel 9-month culturally informed motivational interviewing and electronic messaging intervention- "Cognition After Obstructive Sleep Apnea (OSA) Among Native American People" (CATNAP) to: 1) provide participants with Motivational Interviewing sessions to address obstructive sleep apnea (OSA), positive airway pressure (PAP) adherence, and risk of Alzheimer's disease and related dementias (ADRD) in American Indians and 2) provide participants with electronic messaging to support PAP adherence among American Indian elders, aged 50 years and older.

This study will explore the relationship between OSA and cognitive function and evaluate OSA as a mechanism for the strong association between sleep disorders and Alzheimer's disease and related dementias (ADRD). CATNAP will be implemented as a randomized controlled trial at 4 community sites serving American Indians in the Northern Plains. A total of 300 American Indian elders, aged 50 years and older, with a confirmed OSA diagnosis and prescribed PAP therapy will be randomized to receive usual care consisting of PAP therapy alone (control condition) or usual care plus the culturally informed CATNAP component (intervention condition).

The primary outcome is PAP adherence and secondary outcome cognitive function. The study will partner with Missouri Breaks Industries Research Inc., and Missouri Breaks Durable Medical Equipment to monitor participants PAP use, which is uploaded automatically to the cloud. Outcomes will be measured at baseline, 3-months, and 9-months.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older
* Self report American Indian or Alaskan Native
* diagnosed with obstructive sleep apnea
* prescribed PAP therapy and have a device
* *Ability to understand written and spoken English; and
* *Ability and willingness to follow all study protocols.

Exclusion Criteria:

* Living in a household with someone who is enrolled in the study
* Already using PAP device at Medicaid recommended standards
* Cognitive decline, unable to consent on their own

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Airway Pressure (PAP) minutes per night | 9 months
  Participant mask-on time data collected by the PAP equipment will be extracted as continuous minutes per night.
Nights of PAP use | 9 months
  Proportion of nights with 4+ hours of PAP use from PAP device
PAP adherence | 9-months
  Use of device for more than 240 minutes per night, on 21 or more days out of the past 30 days. From PAP device.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment total score | 9 months
  The Montreal Cognitive Assessment is a widely used self-report instrument to screen for cognitive impairment and probable dementia. It comprises 30 items and takes approximately 10 minutes to complete. The assessment generates a summary score with range of 0 to 30, with scores 25 and above indicating normal cognition. Scores of 19-25 are considered to indicate mild cognitive impairment, scores of 11-21 indicate probable dementia, and scores less than 10 indicating severe cognitive impairment and Alzheimer's disease.
Cognivue total score | 9 months
  The Cognivue Clarity device (Clarity: Comprehensive 10-Minute Cognitive Self Test | Cognivue®) is a 10- to 15-minute patient-administered test that evaluates cognition in 6 domains: visuospatial, executive function, memory, naming/language, delayed recall, and abstraction. Study staff will be present to provide assistance in using the device, as needed. The device generates a summary score with scores 75 and above indicating normal cognitive function, 50-75 indicating mild cognitive impairment, and scores below 50 indicating severe cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Breaks Industries Research Inc, Eagle Butte, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No